CLINICAL TRIAL: NCT03059472
Title: Strong Hearts for New York: A Rural Community CVD Prevention Program
Brief Title: Strong Hearts for New York: A Rural Heart Disease Prevention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Montana State University (Other); Tufts University (Other); Bassett Healthcare (Other); Cornell Cooperative Extension (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB #: 1402004505-2
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Heart Disease; Cardiovascular Disease; Sedentary Lifestyle; Overweight; Obesity
Keywords: physical activity; nutrition; social network; civic engagement
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Sedentary Behavior; Overweight; Obesity; Motor Activity | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Intervention) (Experimental): Full Intervention participants will meet twice per week for one hour each time, for approximately 6 months. Participants will learn and practice good nutrition and physical activity for improved individual, family and community health.
  Interventions: Behavioral: Group 1 (Intervention)
- Group 2 (Delayed intervention) (Experimental): Delayed intervention participants will participate in the same activities as Group 1 but 6 months after Group 1.
  Interventions: Behavioral: Group 2 (Delayed intervention)

INTERVENTIONS:
Behavioral: Group 1 (Intervention) — The investigators will evaluate the efficacy of the SHHC curriculum in a 24-week community-based randomized delayed intervention trial. They will compare changes in CVD-related anthropometric, physiologic, behavioral, and psychosocial parameters between subjects in 5 intervention and 6 delayed intervention communities. In addition, the investigators will evaluate changes in behavior, attitudes, and knowledge among SHHC intervention subjects' "social network".
  Arms: Group 1 (Intervention)
Behavioral: Group 2 (Delayed intervention) — The investigators will evaluate the efficacy of the SHHC curriculum in a 24-week community-based randomized delayed intervention trial. They will compare changes in CVD-related anthropometric, physiologic, behavioral, and psychosocial parameters between subjects in 5 intervention and 6 delayed intervention communities. In addition, the investigators will evaluate changes in behavior, attitudes, and knowledge among SHHC intervention subjects' "social network".
  Arms: Group 2 (Delayed intervention)

SUMMARY:
Strong Hearts for New York is a research study which aims to reduce cardiovascular disease (CVD), improve quality of life, and reduce CVD related health care costs in rural communities. Our aim is to better understand how changes in lifestyle can affect the health of rural women and others in their communities.

DETAILED DESCRIPTION:
There are notable cardiovascular disease (CVD) disparities among people living in rural settings, particularly medically underserved rural areas. Complex factors such as socioeconomic disadvantage, social and cultural dynamics, geographic distances/barriers, and limited access to healthcare, healthy foods, and/or physical activity opportunities contribute to the issue. The objective of Strong Hearts, Healthy Communities (SHHC) is to reduce rural CVD disparities through civic engagement and implementation of a community-based intervention in 11 underserved New York communities. SHHC builds upon a long-standing collaboration with National Institute of Food and Agriculture cooperative extension educators, who will implement the project. There is limited knowledge about how programs and services can move beyond commonly used individual-level approaches-which have limitations in terms of cost, impact, reach, and sustainability-to effectively reduce rural CVD health disparities using an integrated, multi-level, community-engaged approach. The objective of Strong Hearts, Healthy Communities (SHHC) is to address this gap in knowledge and practice by working with residents, practitioners, health educators, local leadership, and other stakeholders in 11 medically underserved rural communities in New York to test a comprehensive program designed to: a) improve diet and physical activity behaviors, b) promote local built environment resources, and c) shift social norms about active living and healthy eating through civic engagement, capacity building, and community based programming.

RANDOMIZED INTERVENTION AND DELAYED INTERVENTION: In the current phase of the project, the efficacy of the SHHC program curriculum will be evaluated in a 24-week delayed intervention trial. The investigators will compare changes in CVD-related anthropometric, physiologic, behavioral, and psychosocial parameters between subjects in 5 intervention and 6 delayed communities in New York State. In addition, changes in behavior, attitudes, and knowledge among SHHC intervention subjects' "social network" will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) greater than or equal to 25
* If BMI is less than 30, not currently physically active
* Blood pressure is less than 160/100 mm Hg
* Heart rate is between 60-100 bpm
* English-speaking
* Able and willing to obtain physician's approval to participate in intervention starting either in March 2017 or September 2017
* Willing to participate in assessment activities
* Willing to make a firm commitment to participate in intervention starting either in Spring or Fall 2017

Exclusion Criteria:

* BMI less than 25
* If BMI is less than 30, currently physically active
* Untreated hypertension
* Heart rate lower than 60 or higher than 100 bpm
* Non-English speaking
* Not able or willing to obtain physician's approval to participate
* Not interested or willing to participate in assessment activities
* Not able or willing to make a firm commitment to participate in intervention starting either in Spring or Fall 2017

Ages: 40 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 182 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline to 24 weeks

SECONDARY OUTCOMES:
Changes in body weight | Baseline to 48 weeks
Changes in blood pressure | Baseline to 24 weeks, 48 weeks
Changes in blood lipids | Baseline to 24 weeks, 48 weeks
Changes in c-reactive protein | Baseline to 24 weeks, 48 weeks
Changes in hemoglobin A1C | Baseline to 24 weeks, 48 weeks
Changes in waist circumference | Baseline to 24 weeks, 48 weeks
Changes in hip circumference | Baseline to 24 weeks, 48 weeks
Changes in 7 day accelerometry | Baseline to 24 weeks, 48 weeks
Changes in 7 day dietary recall | Baseline to 24 weeks, 48 weeks
Changes in healthy eating self-efficacy assessed by questionnaire | Baseline to 24 weeks, 48 weeks
Changes in exercise self-efficacy assessed by questionnaire | Baseline to 24 weeks, 48 weeks
Changes in healthy eating attitudes of social network of participants assessed by questionnaire | Baseline to 24 weeks, 48 weeks
Changes in exercise attitudes of social network of participants assessed by questionnaire | Baseline to 24 weeks, 48 weeks
Changes in healthy eating self-efficacy of social network of participants assessed by questionnaire | Baseline to 24 weeks, 48 weeks
Changes in exercise self-efficacy of social network of participants assessed by questionnaire | Baseline to 24 weeks, 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Seguin, PhD, Principal Investigator — Cornell University
Locations (13):
- United States (13):
  - Clyde, Clyde, New York
  - Cobleskill, Cobleskill, New York
  - Cooperstown, Cooperstown, New York
  - Dolgeville and Little Falls, Dolgeville, New York
  - Hamilton, Hamilton, New York
  - Hartwick, Hartwick, New York
  - Herkimer, Mohawk and Ilion, Herkimer, New York
  - Ithaca, Ithaca, New York
  - Seguin Research Lab, Cornell University, Ithaca, New York
  - Milford, Milford, New York
  - Morrisville, Morrisville, New York
  - Newark, Newark, New York
  - Sharon Springs, Sharon Springs, New York

REFERENCES:
- [Derived] Andreyeva E, Graham ML, Eldridge GD, Folta SC, Nelson ME, Strogatz D, Seguin-Fowler RA. Cost-Effectiveness of Two Iterations of a Community-Based Cardiovascular Disease Prevention Intervention. Obesity (Silver Spring). 2026 Jan;34(1):65-75. doi: 10.1002/oby.70050. Epub 2025 Oct 16. PMID 41102867
- [Derived] Szeszulski J, Rolke LJ, Ayine P, Bailey R, Demment M, Eldridge GD, Folta SC, Graham ML, MacMillan Uribe AL, McNeely A, Nelson ME, Pullyblank K, Rethorst C, Strogatz D, Seguin-Fowler RA. Process evaluation findings from Strong Hearts, Healthy Communities 2.0: a cardiovascular disease prevention intervention for rural women. Int J Behav Nutr Phys Act. 2024 Oct 22;21(1):122. doi: 10.1186/s12966-024-01670-y. PMID 39438920
- [Derived] MacMillan Uribe AL, Demment M, Graham ML, Szeszulski J, Rethorst CD, Githinji P, Nelson ME, Strogatz D, Folta SC, Bailey RL, Davis JN, Seguin-Fowler RA. Improvements in dietary intake, behaviors, and psychosocial measures in a community-randomized cardiovascular disease risk reduction intervention: Strong Hearts, Healthy Communities 2.0. Am J Clin Nutr. 2023 Nov;118(5):1055-1066. doi: 10.1016/j.ajcnut.2023.09.003. Epub 2023 Sep 17. PMID 37717638
- [Derived] Maddock JE, Demment M, Graham M, Folta S, Strogatz D, Nelson M, Ha SY, Eldridge GD, Seguin-Fowler RA. Changes in physical activity outcomes in the Strong Hearts, Healthy Communities (SHHC-2.0) community-based randomized trial. Int J Behav Nutr Phys Act. 2022 Dec 28;19(1):159. doi: 10.1186/s12966-022-01401-1. PMID 36578002
- [Derived] Seguin-Fowler RA, Eldridge GD, Rethorst CD, Graham ML, Demment M, Strogatz D, Folta SC, Maddock JE, Nelson ME, Ha S. Improvements and Maintenance of Clinical and Functional Measures Among Rural Women: Strong Hearts, Healthy Communities-2. 0 Cluster Randomized Trial. Circ Cardiovasc Qual Outcomes. 2022 Nov;15(11):e009333. doi: 10.1161/CIRCOUTCOMES.122.009333. Epub 2022 Nov 15. PMID 36378768
- [Derived] Seguin-Fowler RA, Strogatz D, Graham ML, Eldridge GD, Marshall GA, Folta SC, Pullyblank K, Nelson ME, Paul L. The Strong Hearts, Healthy Communities Program 2.0: An RCT Examining Effects on Simple 7. Am J Prev Med. 2020 Jul;59(1):32-40. doi: 10.1016/j.amepre.2020.01.027. Epub 2020 May 7. PMID 32389532
- [Derived] Pullyblank K, Strogatz D, Folta SC, Paul L, Nelson ME, Graham M, Marshall GA, Eldridge G, Parry SA, Mebust S, Seguin RA. Effects of the Strong Hearts, Healthy Communities Intervention on Functional Fitness of Rural Women. J Rural Health. 2020 Jan;36(1):104-110. doi: 10.1111/jrh.12361. Epub 2019 Mar 13. PMID 30865324